CLINICAL TRIAL: NCT04271631
Title: Integrasi Edukasi Berbasis Aplikasi Dan "CARE Coaching Model" Pada Pengelolaan Pasien Diabetes Mellitus Tipe 2 Yang Menggunakan Insulin
Brief Title: Integration of Education Based-Application and "CARE Coaching Model" in Management of Type 2 Diabetes Mellitus Patients Using Insulin
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Prof. Dr. dr. Pradana Soewondo, SpPD-KEMD, Professor, Endocrinologist, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PS001
Record Dates: First submitted 2020-02-07; First posted 2020-02-17 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Type 2 diabetes mellitus; Mobile Application-Based Diabetes Education; Health Coaching
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Masking Description: Open label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): Received conventional education group
- Intervention 1 (Experimental): Received conventional education group and Mobile Application-Based Diabetes Education
  Interventions: Other: Mobile Application-Based Diabetes Education
- Intervention 2 (Experimental): Received Mobile Application-Based Diabetes Education and Health Coaching
  Interventions: Other: Mobile Application-Based Diabetes Education; Other: Health Coaching

INTERVENTIONS:
Other: Mobile Application-Based Diabetes Education — Additional education was given using application, subjects were asked to open the application at least once a day
  Other Names: DM EduCorner Application
  Arms: Intervention 1; Intervention 2
Other: Health Coaching — Health coaching was given as face to face with a coach
  Arms: Intervention 2

SUMMARY:
Diabetes mellitus is increasing in incidence worldwide. The goal of management of diabetes is to achieve blood sugar control by minimizing side effects and preventing short and long term complications. Self-management becomes important in the management of diabetes mellitus. The use of mobile phone applications provides opportunities for the management of diabetics. In addition, health coaching is one of method used for empowering patients with chronic diseases, such as diabetes. This study aims to evaluate the impact of Mobile Application-Based Diabetes Education and health coaching in management of type 2 diabetes mellitus.

DETAILED DESCRIPTION:
A randomized control trial, pre and post study involving 105 subjects randomized into 3 arms:

* Control : received conventional education group
* Intervention 1 : received conventional education group + mobile application-based diabetes education
* Intervention 2 : received mobile application-based diabetes education + health coaching

Conventional education group divided into 6 session, which for each session consist of 2 different topics and lasts for 60 minutes.

Mobile application-based diabetes education is using DM Educorner (Diabetes Mellitus Education Corner) availablle in Google PlayStore. Education contents was delivered in articles, video and infographics.

Health coaching was given by a coach, a healthcare professional who undergo training to become a coach. Health coaching delivered as face to face between subjects and coach.

Laboratory examination and questionnaire collected at baseline, 3 and 6 months after intervention.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes Mellitus
* multiple daily insulin injection (basal and rapid, or mixed)
* 30 - 65 years old
* HbA1c > 8%
* Using smartphone in daily lives.
* Willing to follow the research by signing an informed consent

Exclusion Criteria:

* Patients with cognitive disease (such as dementia)
* Patients with hearing or sight problem
* Unable to live independently on daily basis
* Patients who have disease that may affect Hba1c such as hemolytic anemia, thalassemia

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2019-06-12 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-05-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Hb1A1c at 3 months | 3 months
  Glycemic control

SECONDARY OUTCOMES:
Change from Baseline Fasting plasma glucose at 3 months | 3 months after intervention
  Glycemic control
Change from Baseline 2 hours-post prandial plasma glucose at 3 months | 3 months after intervention
  Glycemic control
Change from Baseline Total cholesterol at 3 months | 3 months after intervention
  Diabetes Mellitus control
Change from Baseline High-density lipoprotein cholesterol (HDL-c) at 3 months | 3 months after intervention
  Diabetes Mellitus control
Change from Baseline Low-density lipoprotein cholesterol (LDL-c) at 3 months | 3 months after intervention
  Diabetes Mellitus control
Change from Baseline Triglycerides at 3 months | 3 months after intervention
  Diabetes Mellitus control
Mean of intake calories from food Record | at baseline, 3 months after intervention
  mean calorief from diet intake in 3 days
Global Physical Activities Questionnaire | at baseline, 3 and 6 months after intervention
  Questionnaire about physical activities in whole one week. Divided into 3 categories: low, moderate, high. Every categories describe duration and numbers of day being active during 1 weeks and not for judging it is good or worse.
Self-Monitoring Blood Glucose | through study completion, an average of 3 months
  Notes of daily blood glucose

CONTACTS AND LOCATIONS:
Overall Officials: Pradana Soewondo, Prof, Principal Investigator — Fakultas Kedokteran Universitas Indonesia
Locations (1):
- Faculty of Medicine, Universitas Indonesia, Jakarta Pusat, DKI Jakarta, Indonesia